CLINICAL TRIAL: NCT00643266
Title: Memory Interventions for Older Adults
Brief Title: Recollection Training in Healthy Older Adults and Older Adults With Amnestic Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Nicole D. Anderson, Senior Scientist, Baycrest
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RecollectionTraining; CIHR MOP 67015; ASC 08 95
Record Dates: First submitted 2008-02-26; First posted 2008-03-26 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Amnestic Mild Cognitive Impairment; Aging
Keywords: recollection training; aging; amnestic mild cognitive impairment; fMRI
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Recollection training via graduated increases in task difficulty, carried out over 36 sessions over 9 training days
  Interventions: Behavioral: Recollection Training
- 2 (Active Comparator): Computer-delivered information sessions about memory and aging with Jeopardy-like games to engage participants
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Recollection Training — Participants are exposed to long lists of words. Each word is presented either visually or auditorily, and each word is repeated after a variable number of intervening words (the lag), in each the same modality, or the other modality. Participants are instructed to respond "yes" only to words repeated in the same modality. If a performance criterion is met, the lag is increased for the next session; if the performance criterion is not met, the same lag is repeated in the next session.
  Other Names: Memory training
  Arms: 1
Behavioral: Control — Participants view PowerPoint presentations on various topics related to memory and aging (e.g., structural brain changes, diet, stress, depression) and how each of these topics affect memory, and after each presentation, play a Jeopardy-like game to test their knowledge gain
  Other Names: Educational Control
  Arms: 2

SUMMARY:
We have developed a training intervention that successfully improves older adults' memory. We have also shown that older adults whose memory is as good as younger adults' memory (Hi-Old) use an altered pattern of memory-related brain activity compared to younger adults, whereas healthy older adults with poorer memory (Lo-Old) do not. We have also shown that individuals with amnestic Mild Cognitive Impairment (aMCI) have impairments of conscious, effortful, Recollection-based memory processes, whereas their automatic, Familiarity-based memory processes are intact. Our primary current goal is to investigate whether our successful memory intervention will improve Recollection and produce induce altered patterns of brain activity in the Lo-Old and aMCI.

Young, Lo-Old, Hi-Old, and aMCI will be scanned using functional magnetic resonance imaging while performing two memory tasks. Half of the Lo-Old and half of the aMCI will then receive the memory intervention, while the other half in each group will receive a control program consisting of information and games about aging. The Lo-Old and aMCI will then be rescanned while performing the two memory tasks. We predict that the memory intervention will improve performance on a number of memory tasks, and will induce altered patterns of brain activity. In the Lo-Old, their brain activity after the memory intervention will look more like the Hi-Old, while brain activity will become more focal in the aMCI.

ELIGIBILITY:
Inclusion Criteria:

* 65-90 years old
* English as a first language or learned before kindergarten
* Right handed

Exclusion Criteria:

* Neurologic disorder
* Major medical disorder affecting cognition
* Psychiatric disorder
* Metal in the body that poses a hazard in the MRI scanner

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Recollection estimates | Immediately post-training and three months post-training
  Recollection, defined as Correct "yes" responses to "Same" repetitions minus Incorrect "yes" responses to "Different" repetitions, as a function of condition (trained versus control), lag (3, 16) and time (pre-, post-, and 3 month follow-up)

SECONDARY OUTCOMES:
Brain activation as assessed by functional magnetic resonance imaging | Immediately post-training
  Prefrontal (inferior, middle, and superior frontal gyri) activation for Different Repetitions minus Same Repetitions, as a function of group (trained versus control), lag (3, 16), and time (pre, post). Additional analyses will compare trained versus control older adults with younger adults on these measures at baseline (pre). Analyses will include an exploration of prefrontal laterality of the effects (left minus right), to see whether training induces greater bilaterality of activation.
Transfer to other recollection-dependent task and to subjective memory measures | Immediately post-training and three months post-training
  Source memory, self-ordered pointing, n-back, a Sternberg task, CVLT, an AB-AC test of proactive interference, the Memory Controllability Inventory, Multifactorial Memory Questionnaire (Ability and Contentment subscales), Meta-Memory in Adulthood questionnaire (locus of control, anxiety, and capability subscales), and an in-house measure of the efficacy of the control program

CONTACTS AND LOCATIONS:
Overall Officials: Nicole D Anderson, PhD, CPsych, Principal Investigator — Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

REFERENCES:
- [Result] Anderson ND, Ebert PL, Jennings JM, Grady CL, Cabeza R, Graham SJ. Recollection- and familiarity-based memory in healthy aging and amnestic mild cognitive impairment. Neuropsychology. 2008 Mar;22(2):177-87. doi: 10.1037/0894-4105.22.2.177. PMID 18331160
- [Result] Guild EB, Vasquez BP, Maione AM, Mah L, Ween J, Anderson ND. Dynamic working memory performance in individuals with single-domain amnestic mild cognitive impairment. J Clin Exp Neuropsychol. 2014;36(7):751-60. doi: 10.1080/13803395.2014.941790. Epub 2014 Aug 30. PMID 25175752
- [Result] Ebert PL, Anderson ND. Proactive and retroactive interference in young adults, healthy older adults, and older adults with amnestic mild cognitive impairment. J Int Neuropsychol Soc. 2009 Jan;15(1):83-93. doi: 10.1017/S1355617708090115. PMID 19128531
- [Result] Anderson ND, Ebert PL, Grady CL, Jennings JM. Repetition lag training eliminates age-related recollection deficits (and gains are maintained after three months) but does not transfer: Implications for the fractionation of recollection. Psychol Aging. 2018 Feb;33(1):93-108. doi: 10.1037/pag0000214. PMID 29494181
- [Result] Meusel LA, Grady CL, Ebert PE, Anderson ND. Brain-behavior relationships in source memory: Effects of age and memory ability. Cortex. 2017 Jun;91:221-233. doi: 10.1016/j.cortex.2016.12.023. Epub 2017 Jan 12. PMID 28161030